CLINICAL TRIAL: NCT00005854
Title: Transplantation of HLA Haploidentical Marrow Cells After Ex Vivo Exposure to Recipient Alloantigen in Presence of CTLA4-Ig - A Phase II Study of Tolerance Induction in Donor T Cells by Blockade of the CD80/CD86:CD28 Costimulatory Signal
Brief Title: Bone Marrow Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1457.00; FHCRC-1457.00; NCI-H00-0059; CDR0000067879 (Registry Identifier: PDQ)
Record Dates: First submitted 2000-06-02; First posted 2004-06-28 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: recurrent childhood acute lymphoblastic leukemia; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Cyclophosphamide; Cyclosporine; Methotrexate; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation
Procedure: in vitro-treated bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy and radiation therapy used to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of bone marrow transplantation in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the incidence and severity of acute graft versus host disease after transplantation of HLA haploidentical bone marrow preincubated with alloantigen and CTLA4-Ig ex vivo in patients with hematologic malignancies. II. Determine the engraftment rate with this treatment regimen in these patients. III. Determine the safety of this treatment regimen in these patients. IV. Determine the incidence of infection and relapse after this treatment regimen in these patients. V. Determine whether host specific tolerance develops in these patients after receiving this treatment regimen.

OUTLINE: This is a multicenter study. Patients undergo leukapheresis to collect white blood cells which are incubated with donor bone marrow cells in the presence of CTLA4-Ig for 36 hours. Patients undergo total body irradiation on days -7, -6, -5, and -4 and receive cyclophosphamide IV on days -3 and -2. Patients with acute lymphocytic leukemia, prior lymphoid blast crisis chronic myelogenous leukemia, high grade non-Hodgkin's leukemia (NHL), intermediate grade NHL with prior marrow or extramedullary disease, or prior CNS leukemia receive 2 doses of methotrexate intrathecally prior to bone marrow transplantation, and 4-6 doses following. Patients receive bone marrow transplantation on day 0; methotrexate IV on days 1, 3, 6, and 11; and cyclosporine IV on days -1 to 50. Patients are followed weekly for 1 month, monthly for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study over 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Any of the following hematologic malignancies: Acute myelogenous leukemia in second or greater remission or relapse High risk acute lymphoblastic leukemia First complete remission with high risk cytogenetics [e.g., t(9;22), t(8;14), or t(4;11)] or slow early response OR Any second or greater remission OR Relapse or induction failure Relapsed non-Hodgkin's lymphoma (NHL) with chemotherapy sensitive disease Multiple myeloma with chemotherapy sensitive disease Chronic lymphocytic leukemia with chemotherapy sensitive disease Myelodysplastic syndrome Chronic myelogenous leukemia (CML) in accelerated phase, blast phase, or remission after blast phase Juvenile CML Patients must have haploidentical donors and meet the following criteria: Lack an HLA A, B, and DR matched related donor Lack an HLA A, B, DRB1 matched or single allele mismatched unrelated donor or for whom the following apply: High likelihood of rapid disease progression while an unrelated donor search is in progress AND Review of the patient HLA typing, gene frequency, results of the preliminary search and the donor pool suggest that a donor will not be found within a suitable time frame Lack an HLA A, B, DRB1 matched cord blood unit or lack a cord blood unit that has an adequate cell dose and is mismatched for 1-2 HLA A, B, DRB1 Do not have an indication for autologous transplant, including patients with NHL or multiple myeloma who are not eligible for autologous transplant Negative antidonor antibody crossmatch

PATIENT CHARACTERISTICS: Age: Under 51 Performance status: Not specified Life expectancy: No patients with life expectancy severely limited by diseases other than malignancy Hematopoietic: See Disease Characteristics Hepatic: AST no greater than 2 times normal Renal: Creatinine no greater than 2 times normal OR Creatinine clearance at least 50% for age, weight, and height Cardiovascular: No cardiac insufficiency requiring treatment No symptomatic coronary artery disease Pulmonary: No severe hypoxemia pO2 less than 70 mm Hg with decreased DLCO less than 70% predicted OR No mild hypoxemia pO2 less than 80 mm Hg with severely decreased DLCO less than 60% predicted Other: HIV negative Not pregnant or nursing Fertile patients must use effective contraception during and for one year after study No leukoencephalopathy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No more than 3,000 cGy prior radiotherapy to brain No more than 1,500 cGy prior radiotherapy to chest or abdomen Surgery: Not specified

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1999-12; Study Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann E. Woolfrey, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (4):
- United States (4):
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of South Carolina School of Medicine, Columbia, South Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington